CLINICAL TRIAL: NCT01020838
Title: An Open-label, Non-randomized Study to Evaluate the Efficacy and Safety of BAY94-9172 (ZK 6013443) Positron Emission Tomography (PET) Imaging for Detection/Exclusion of Cerebral Beta-amyloid When Compared to Postmortem Histopathology
Brief Title: Phase III Study of Florbetaben (BAY94-9172) PET Imaging for Detection/Exclusion of Cerebral β-amyloid Compared to Histopathology
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Life Molecular Imaging SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14595; 2009-012569-79 (EudraCT Number)
Record Dates: First submitted 2009-11-16; First posted 2009-11-26 (Estimated); Results first posted 2015-03-25 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-04

CONDITIONS: Alzheimer Disease
Keywords: Florbetaben; Amyloid beta-protein; Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease; Plaque, Amyloid | interventions — 4-(N-methylamino)-4'-(2-(2-(2-fluoroethoxy)ethoxy)ethoxy)stilbene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Florbetaben (BAY94-9172) (Experimental)
  Interventions: Drug: Florbetaben (BAY94-9172)

INTERVENTIONS:
Drug: Florbetaben (BAY94-9172) — Single intravenous injection 1-5ml, 300 MBq (+/- 20%)

SUMMARY:
To determine the sensitivity and specificity of the visual assessment of tracer uptake in the Florbetaben PET images compared to histological verification of the presence or absence of cerebral β-amyloid in the respective histopathologic post mortem specimens as the standard of truth

ELIGIBILITY:
Inclusion Criteria:

* Females, no child-bearing potential or negative urine pregnancy test on day of BAY94-9172 injection
* Exhibits visual, auditory, and communicative capabilities adequate to provide informed consent or assent and comply with study procedures
* Is willing and able to lie down in magnetic resonance imaging (MRI) and positron emission tomography (PET) scanners
* Is willing to donate their brain for postmortem examination in case of death
* The subject, or the subject and/or legally acceptable representative will be compliant and have a high probability of completing the study in the opinion of the investigator
* Has been fully informed about the study, including provisions of the Health Insurance Portability and Accountability Act (HIPAA), as applicable, and informed consent or assent has been signed and dated (with time) by the subject and/or the subject's legally acceptable representative
* The subjects who have participated in a previous florbetaben study e.g. study 311741 may be included in the present study. The MRI- and florbetaben PET scan do not need to be repeated if both scans were performed within twelve months prior to inclusion.

Exclusion Criteria:

* Has severe cerebral macrovascular (ie, multi-stroke) disease or brain tumor (metastasis/brain cancer) as verified by MRI
* Has any contraindication to magnetic resonance imaging (MRI) examination, eg, metal implants or phobia as determined by the onsite radiologist performing the scan
* Has been previously enrolled in this study or participated in a clinical study involving an investigational pharmaceutical product within 30 days prior to screening and/or was administered a radiopharmaceutical within 10 radioactive half-lives prior to study drug administration in this study
* Has severe cardio-vascular instability requiring intensive care surveillance and/or therapeutic intervention (i.e. catecholamine infusion)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2009-11; Primary Completion 2011-09 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Piramal Imaging SA Study Director, Study Director — Life Molecular Imaging SA
Locations (17):
- United States (8):
  - Sun City, Arizona
  - Stanford, California
  - Tampa, Florida
  - Teaneck, New Jersey
  - Philadelphia, Pennsylvania
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
- Heidelberg, Victoria, Australia
- France (2):
  - Lille
  - Strasbourg
- Germany (2):
  - Jülich, North Rhine-Westphalia
  - Leipzig, Saxony
- Japan (4):
  - Toyohashi, Aichi-ken
  - Isesaki, Gunma
  - Hamamatsu, Shizuoka
  - Itabashi-ku, Tokyo

REFERENCES:
- [Derived] Seibyl J, Catafau AM, Barthel H, Ishii K, Rowe CC, Leverenz JB, Ghetti B, Ironside JW, Takao M, Akatsu H, Murayama S, Bullich S, Mueller A, Koglin N, Schulz-Schaeffer WJ, Hoffmann A, Sabbagh MN, Stephens AW, Sabri O. Impact of Training Method on the Robustness of the Visual Assessment of 18F-Florbetaben PET Scans: Results from a Phase-3 Study. J Nucl Med. 2016 Jun;57(6):900-6. doi: 10.2967/jnumed.115.161927. Epub 2016 Jan 28. PMID 26823561
- [Derived] Sabri O, Sabbagh MN, Seibyl J, Barthel H, Akatsu H, Ouchi Y, Senda K, Murayama S, Ishii K, Takao M, Beach TG, Rowe CC, Leverenz JB, Ghetti B, Ironside JW, Catafau AM, Stephens AW, Mueller A, Koglin N, Hoffmann A, Roth K, Reininger C, Schulz-Schaeffer WJ; Florbetaben Phase 3 Study Group. Florbetaben PET imaging to detect amyloid beta plaques in Alzheimer's disease: phase 3 study. Alzheimers Dement. 2015 Aug;11(8):964-74. doi: 10.1016/j.jalz.2015.02.004. Epub 2015 Mar 28. PMID 25824567

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened at 15 study centers in Australia, Germany, France, Japan, and the U.S.
Groups:
- All Study Participants: All patients enrolling into the study
Period: Overall Study
Arm/Group | All Study Participants
Started | 218
Safety Analysis Set | 216 (Two patients were excluded from this population because injection of florbetaben was not done.)
Interim Analysis Set (Primary Efficacy) | 41 (Primary efficacy analysis of initial study period (tissue-scan matched regional analysis))
Final Analysis Set (Whole Brain) | 97 (Final analysis set comparing PET scans with different histopathological evaluations.)
First Annual Repeat Injection | 91 (Patients returning for first follow-up administration and PET-scan.)
Second Annual Repeat Injection | 34 (Patients returning for second follow-up administration and PET-scan.)
Completed | 35
Not Completed | 183
Not completed — Death | 90
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 9
Not completed — Lost to Follow-up | 6
Not completed — Most common: Study ended by sponsor | 77

BASELINE CHARACTERISTICS:
Population: Participants in the safety analysis set were treated with study drug.
Groups:
- Safety Analysis Set: All study participants who received any amount of florbetaben were included in the safety analysis set.
Arm/Group | Safety Analysis Set
Number analyzed (Participants) | 216
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.4 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104
  Male | 112
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 213
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 55
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 159
  More than one race | 0
  Unknown or Not Reported | 0
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 23.617 (5.213)
Body weight [Mean (Standard Deviation); unit: kg] | 64.95 (18.44)
Height [Mean (Standard Deviation); unit: cm] | 164.70 (12.34)
Baseline clinical diagnosis [Number; unit: participants]
  Alzheimer's Disease | 137
  Dementia with Lewy bodies | 5
  Other dementia subject | 31
  Healthy volunteers | 32
  Healthy negative control | 11

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity and Specificity of the Majority Read of Visual Assessment of Tracer Uptake Compared to Histological Verification of the Presence or Absence of Cerebral Beta-amyloid in Postmortem Specimens
Description: The sensitivity/specificity of the visual assessment were calculated based on the majority read assessment of regional tracer uptake. This result was derived from assessments by 3 independent readers for brain regions of a subject where a Standard of Truth (SOT) was available. The SOT for this analysis was a centralized histopathological determination of β-amyloid presence/absence based on both Bielschowsky silver and immunohistochemical staining. Based on the PET images, a brain region was classified as "normal" or "abnormal" depending on the presence or absence of regional tracer uptake in the respective region. "Normal" therefore meant absence of β-amyloid and "abnormal" presence of β-amyloid. Sensitivity was defined as the percentage of abnormal brain regions from all regions where an SOT was available and the SOT was "β-amyloid present". Specificity was defined as the percentage of normal brain regions from all regions where an SOT was available and was "β-amyloid not present".
Time Frame: 90-110 minutes post injection (PET image acquisition)
Population: All participants included in the Interim Analysis Set were included in this analysis.
Measure: Number; unit: percentage of regions
Groups:
- Sensitivity (Interim Analysis Set); Specificity (Interim Analysis Set): The full analysis set consisted of 31 subjects for whom both brain specimen with a valid Standard of Truth (SOT) in at least one brain region and a florbetaben PET scan were available and 10 healthy controls for whom a florbetaben PET scan was available and whose SOT was considered β-amyloid negative by definition.
Arm/Group | Sensitivity (Interim Analysis Set) | Specificity (Interim Analysis Set)
Number analyzed (Participants) | 41 | 41
percentage of regions
  Total | 77.36 | 94.20
  Frontal Cortex | 85.71 | 95.00
  Occipital Cortex | 88.89 | 86.36
  Hippocampus | 57.14 | 100.00
  Anterior Cingulate Cortex | 90.00 | 85.71
  Posterior Cingulate Cortex | 81.82 | 94.44
  Cerebellar Cortex | 0.00 | 100.00
Statistical Analysis 1: Comparison: Sensitivity (Interim Analysis Set); For the primary analysis, point estimates together with normal-approximated, two sided 95% confidence intervals, were given for sensitivity in beta-amyloid detection based on the majority read. The following hypothesis was formulated for sensitivity: H0,sens: sensitivity ≤ 0.6 vs. H1, sens: sensitivity > 0.6 H0,sens was to be rejected if the lower bound of the two-sided 95% CI is larger than 0.6; Test type: Superiority or Other; Sensitivity = 0.774, 95% CI 2-sided [0.654 to 0.894] — Point estimate of sensitivity was calculated by the method of Rao and Scott. Variance for sensitivity is based on subjects that contribute at least one brain region, which is amyloid positive according to the SoT
Statistical Analysis 2: Comparison: Specificity (Interim Analysis Set); For the primary analysis, point estimates together with normal-approximated, two sided 95% confidence intervals, were given for specificity in amyloid detection based on the majority read. The following hypothesis was formulated for specificity: H0,spec: specificity ≤ 0.8 vs. H1, spec: specificity > 0.8 H0,spec was to be rejected if the lower bound of the two-sided 95% CI is larger than 0.8; Test type: Superiority or Other; Specificity = 0.942, 95% CI 2-sided [0.886 to 0.998] — Point estimate of specificity was calculated using the method of Rao and Scott. Variance for specificity is based on subjects that contribute at least one brain region, which is amyloid negative according to the SoT

2. Secondary Outcome: Sensitivity and Specificity of the Majority Read "Whole Brain" Visual Assessment in Detecting/Excluding Cerebral Neuritic β-amyloid Plaques Compared With the Histopathological Verification With Bielschowsky Silver Staining (SOT 1).
Description: Sensitivity and specificity of the whole brain visual assessment were calculated. Any brain with a region classified as abnormal from PET imaging was to be classified as abnormal for the "whole brain" assessment. This result was derived from assessments by 3 independent readers for a subject where a Standard of Truth (SOT) was available. The SOT for this analysis was based on a centralized histopathological assessment of the presence/absence of β-amyloid based on Bielschowsky silver staining (SOT 1).
  The sensitivity was defined as the proportion of brains classified as abnormal from all brains where this SOT was available and was "β-amyloid present". The specificity was defined as the proportion of brains classified as normal from all brains where this SOT was available and was "β-amyloid not present".
Time Frame: 90-110 minutes post injection (PET image acquisition)
Population: Sensitivity and Specificity of the Majority Read "Whole Brain" Visual Assessment in Detecting/Excluding Cerebral β-amyloid Plaques Compared with the Histopathological Verification with Bielschowsky silver staining (SOT 1).
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- Full Analysis Set Final Clinical Study Report: The full analysis of the final clinical study report consisted of data from 97 subjects, including 87 subjects with brain specimens and 10 young healthy controls considered to be β-amyloid-negative as a valid Standard of Truth (SOT).
Arm/Group | Full Analysis Set Final Clinical Study Report
Number analyzed (Participants) | 97
percentage of subjects
  Sensitivity | 96.49 [91.71 to 100.00]
  Specificity | 85.00 [73.93 to 96.07]

3. Secondary Outcome: Sensitivity and Specificity of the Majority Read "Whole Brain" Visual Assessment in Detecting/Excluding Cerebral Neuritic β-amyloid Plaques Compared With Histopathological Verification With Bielschowsky Silver Staining and Immunohistochemistry (SOT 2).
Description: Sensitivity and specificity of the whole brain visual assessment were calculated. Any brain with a region classified as abnormal from PET imaging was to be classified as abnormal for the "whole brain" assessment. This result was derived from assessments by 3 independent readers for a subject where a Standard of Truth (SOT) was available. The SOT for this analysis was based on a centralized histopathological assessment of the presence/absence of β-amyloid based on Bielschowsky silver staining and immunohistochemistry (SOT 2).
  The sensitivity was defined as the proportion of brains classified as abnormal from all brains where this SOT was available and was "β-amyloid present". The specificity was defined as the proportion of brains classified as normal from all brains where this SOT was available and was "β-amyloid not present".
Time Frame: 90-110 minutes post injection (PET image acquisition)
Population: Sensitivity and Specificity of the Majority Read "Whole Brain" Visual Assessment in Detecting/Excluding Cerebral neuritic β-amyloid Plaques Compared with the Histopathological Verification with Bielschowsky silver staining and immunohistochemistry (SOT 2).
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Full Analysis Set Final Clinical Study Report
Number analyzed (Participants) | 97
percentage of subjects
  Sensitivity | 96.72 [92.25 to 100.00]
  Specificity | 94.44 [86.96 to 100.00]

4. Secondary Outcome: Sensitivity and Specificity of the Majority Read "Whole Brain" Visual Assessment in Detecting/Excluding Cerebral Neuritic β-amyloid Plaques Compared With the Histopathological Verification According to CERAD Criteria (SOT 3).
Description: Sensitivity and specificity of the whole brain visual assessment were calculated. Any brain with a region classified as abnormal from PET imaging was to be classified as abnormal for the "whole brain" assessment. This result was derived from assessments by 3 independent readers for a subject where a Standard of Truth (SOT) was available. The SOT for this analysis was based on a histopathological assessment of the presence/absence of β-amyloid according to CERAD Criteria (SOT 3).
  The sensitivity was defined as the proportion of brains classified as abnormal from all brains where this SOT was available and was "β-amyloid present". The specificity was defined as the proportion of brains classified as normal from all brains where this SOT was available and was "β-amyloid not present".
Time Frame: 90-110 minutes post injection (PET image acquisition)
Population: Sensitivity and Specificity of the Majority Read "Whole Brain" Visual Assessment in Detecting/Excluding Cerebral β-amyloid Plaques Compared with the Histopathological Verification according to CERAD Criteria (SOT 3).
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Full Analysis Set Final Clinical Study Report
Number analyzed (Participants) | 97
percentage of subjects
  Sensitivity | 96.49 [91.71 to 100.00]
  Specificity | 85.00 [73.93 to 96.07]

5. Secondary Outcome: Sensitivity and Specificity of the Subject Level Composite SUVR Calculated Based on Pathology Results.
Description: Sensitivity and specificity of subject level composite Standard Uptake Value Ratios (SUVR) by SOT for subjects with available brain tissue and 10 healthy volunteers. The SUVR were determined as a quantitative measure of tracer uptake. The SUV is defined as the ratio of the tissue radioactivity concentration c (in MBq/kg) at time point t, and the injected activity (in MBq), extrapolated to the same time (t) divided by the body weight (in kg). SUV numbers were then used to derive SUV ratios (SUVR) using the SUV from the cerebellar cortex as reference. SOTs comprised Bielschowsky silver staining (SOT 1), Bielschowsky silver staining with immunohistochemistry (SOT 2) and neuropathology assessment according to CERAD (SOT 3). SUVR analysis was performed for baseline and available follow-up scans. The optimal threshold for the distinction between β-amyloid present yes/no according to the respective SOT was derived based on ROC curve analyses and used to calculate sensitivity and specificity.
Time Frame: 90-110 minutes post injection (PET image acquisition)
Population: Sensitivity and Specificity of the subject level Composite SUVR with three different SOTs.
Measure: Number; unit: percentage of subjects
Groups:
- Sensitivity of Subject Level Composite SUVR by SOT: The analysis set consisted of data from 96 subjects, including 86 subjects with brain specimens and 10 young healthy controls considered to be β-amyloid-negative as a valid Standard of Truth (SOT). Sensitivity of subject level composite SUVR by SOT for baseline scans and last available scans are reported.
- Specificity of Subject Level Composite SUVR by SOT: The analysis set consisted of data from 96 subjects, including 86 subjects with brain specimens and 10 young healthy controls considered to be β-amyloid-negative as a valid Standard of Truth (SOT). Specificity of subject level composite SUVR by SOT for baseline scans and last available scans are reported.
Arm/Group | Sensitivity of Subject Level Composite SUVR by SOT | Specificity of Subject Level Composite SUVR by SOT
Number analyzed (Participants) | 96 | 96
percentage of subjects
  SOT 1 (initial period) | 89 | 82
  SOT 2 (initial period) | 90 | 91
  SOT 3 (initial period) | 89 | 90
  SOT 1 (last available scan) | 88 | 85
  SOT 2 (last available scan) | 89 | 94
  SOT 3 (last available scan) | 95 | 87

6. Secondary Outcome: Subject Level Composite SUVRs by SOT for Baseline and Available Follow-Up Scans
Description: Subject level composite SUVRs (calculated as mean of SUVRs from the frontal, parietal, lateral temporal, anterior and posterior cingulate, and occipital cortices) by SOT are reported for subjects with available brain tissue. The initial drug administration group includes additionally 10 healthy controls who were considered as ß-amyloid negative. The SOTs for deceased subjects were based on Bielschowsky silver staining (SOT 1), Bielschowsky silver staining in combination with immunohistochemistry (SOT 2) and neuropathology assessment according to CERAD (SOT 3). SUVR analysis was performed for baseline and available follow-up scans.
Time Frame: 90-110 minutes post injection (PET image acquisition)
Measure: Mean (Standard Deviation); unit: Standardized Uptake Value Ratio (SUVR)
Groups:
- Initial Drug Administration: The analysis set consisted of data from 96 subjects, including 86 subjects with brain specimens and 10 young healthy controls considered to be β-amyloid-negative as a valid Standard of Truth (SOT). Descriptive statistics of subject level Composite SUVR by SOT for baseline scans and last available scans are reported.
- 1st Repeat Drug Administration: The analysis set consisted of data from 20 subjects with brain specimens available.
- 2nd Repeat Drug Administration: The analysis set consisted of data from 3 subjects with brain specimens available.
Arm/Group | Initial Drug Administration | 1st Repeat Drug Administration | 2nd Repeat Drug Administration
Number analyzed (Participants) | 96 | 20 | 3
Standardized Uptake Value Ratio (SUVR)
  SOT 1 (abeta absent) | 1.296 (0.232) | 1.319 (0.414) | 1.537 (NA) — Sample size too low
  SOT 1 (abeta present) | 1.707 (0.276) | 1.625 (0.250) | 1.699 (0.046)
  SOT 2 (abeta absent) | 1.237 (0.140) | 1.175 (0.364) | 1.537 (NA) — Sample size too low
  SOT 2 (abeta present) | 1.714 (0.273) | 1.632 (0.244) | 1.699 (0.046)
  SOT 3 (abeta absent) | 1.263 (0.170) | 1.260 (0.390) | NA (NA) — Sample size too low
  SOT 3 (abeta present) | 1.729 (0.270) | 1.639 (0.236) | 1.645 (0.099)

ADVERSE EVENTS:
Time Frame: All treatment emergent adverse events were recorded within 7 days of the application or follow-up application of study drug.
Description: As this study was conducted in an end-of-life population, death occurring outside 7 day follow-up period after administration of the drug was not collected as part of the study SAE data unless investigator considered the event to be related to drug administration or study procedure.
Groups:
- Initial Drug Administration: Subjects with TEAEs within 7 days of the initial administration of florbetaben.
- 1st Repeat Drug Administration: Subjects with TEAEs within 7 days of the 1st repeat drug administration.
- 2nd Repeat Drug Administration: Subjects with TEAEs within 7 days of the 2nd repeat drug administration.
Arm/Group | Initial Drug Administration | 1st Repeat Drug Administration | 2nd Repeat Drug Administration
Serious Adverse Events (participants affected / at risk) | 12/216 | 0/91 | 0/34
Other Adverse Events (participants affected / at risk) | 48/216 | 22/91 | 14/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Initial Drug Administration (N=216) | 1st Repeat Drug Administration (N=91) | 2nd Repeat Drug Administration (N=34)
Frontotemporal dementia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dementia, Alzheimers' type (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pubis fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Colon cancer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hepatic cancer metastatic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Heat stroke (General disorders) | 1 (1) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac Failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Initial Drug Administration (N=216) | 1st Repeat Drug Administration (N=91) | 2nd Repeat Drug Administration (N=34)
Injection site erythema (General disorders) | 4 (4) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 4 (4) | 0 (0) | 0 (0)
Puncture site reaction (General disorders) | 7 (7) | 4 (4) | 0 (0)
Pyrexia (General disorders) | 7 (8) | 2 (2) | 0 (0)
Blood pressure increased (Investigations) | 3 (3) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 5 (5) | 1 (1) | 1 (1)
Injection site hematoma (General disorders) | 10 (10) | 1 (1) | 0 (0)
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 1 (1)
Haematoma (Vascular disorders) | 1 (1) | 5 (5) | 6 (6)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (5) | 3 (3)
Injection site hemorrhage (General disorders) | 1 (1) | 4 (4) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1) | 0 (0)
Injection site bruising (General disorders) | 5 (5) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 0 (0) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Vessel puncture site swelling (General disorders) | 1 (1) | 1 (1) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Procedural hypertension (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less